CLINICAL TRIAL: NCT03275337
Title: Cerebellar Neuromodulation to Enhance Fear Extinction and Predict Response to Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017_001_01
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorders; Social Phobia
Keywords: Social Phobia; Anxiety; Cerebellum; tDCS; Neuromodulation; Fear Extinction
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Anodal tDCS (Experimental): Anodal tDCS will be performed over bilateral cerebellar hemispheres for 20-minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- Cathodal tDCS (Experimental): Cathodal tDCS will be performed over bilateral cerebellar hemispheres for 20-minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Active Comparator): Sham tDCS will be performed over bilateral cerebellar hemispheres for 20-minutes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS is a non-invasive form of neuromodulation in which direct current is administered placed over a brain region of interest to induce physiological changes such as inhibition or excitation over that region.
  Other Names: tDCS

SUMMARY:
Emerging neuroimaging studies have shown that the cerebellum contributes to different aspects of timing, prediction, learning, and extinction of conditioned responses to aversive stimuli, factors that may be relevant to the success of exposure based behavioral therapy. Our goals are to determine the cerebellar contributions to fear extinction by attempting to modulate key pathways in this process by theta burst stimulation. The long term goal is to lay the foundation for future studies in which neuromodulation is used to augment exposure therapy.

DETAILED DESCRIPTION:
Participants in this study will undergo an assessment for past history and present symptoms of mood, anxiety, trauma, substance abuse, and eating disorders. Safety screening for functional MRI (fMRI) and repetitive transcranial magnetic stimulation (rTMS) will be performed prior to enrollment.

Phase 1 of the study involves two visits. The first visit involves undergoing an fMRI scan and a motor thresholding procedure for rTMS. A clinical assessment will be performed for the above symptoms, or a recap of symptoms if the participant had been previously assessed at our institute.

The second visit involves a fear conditioning session performed in the fMRI scanner followed by one session of rTMS over either a cerebellar or occipital lobe (control) target. This will be immediately followed by a fear extinction phase, also in the fMRI scanner. The participant will return in 24hours to determine consolidation of the fear extinction process.

Phase 2 is similar to Phase 1, except that each participant will undergo two sessions of the fear conditioning and fear extinction phases while undergoing an fMRI scan. In one session, they will receive rTMS over a cerebellar target. In the other session, they will receive rTMS over a control site. These sessions will be separated by at least 1 week.

The participants will then undergo 10 weeks of exposure therapy for social phobia. The goal is to determine whether neuroplasticity related to cerebellar stimulation can predict the response to exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Generalize Anxiety or Social Phobia with an OASIS score =>8

Exclusion Criteria:

* Safety concerns related to undergoing an fMRI scan or tDCS, such as metal in the head, history of unprovoked seizures in self or a first-degree family member, medications that reduce seizure threshold, pregnant or planning to become pregnant.
* History of Post Traumatic Stress Disorder, Obsessive Compulsive Disorder, Panic Disorder, Current Major Depressive Illness, Substance Abuse in the past 1-year, or any thought disorder such as schizophrenia or bipolar disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Activation of ventromedial prefrontal cortex after cerebellar stimulation | Phase 1, Years 1-3
  Activation of vmPFC

SECONDARY OUTCOMES:
Change in resting state connectivity between vmPFC and cerebellar stimulation target | Phase 1, Years 1-3
  Change in resting state connectivity between vmPFC and cerebellum after cerebellar stimulation
Baseline cerebellar-cerebral connectivity prediction of exposure therapy outcomes | Phase 2, Years 3-5
  Baseline cerebellar-cerebral connectivity prediction of exposure therapy outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Hee Cha, MD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No